CLINICAL TRIAL: NCT02039258
Title: A Single-Dose, Open-Label, Randomized, 2-Period Crossover Study to Assess the Effect of Food Coadministration on the Pharmacokinetics of a Fixed Dose Combination Tablet of Canagliflozin (JNJ-28431754) and Metformin Extended Release in Healthy Subjects
Brief Title: Pharmacokinetics of a Fixed Dose Combination of Canagliflozin/Metformin Coadministered With Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR103259; 28431754DIA1064 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Canagliflozin; Metformin; INVOKANA®; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence AB (Experimental): A single dose of CANA/MET XR FDC tablet of 150 mg/1,000 mg under fasted conditions (treatment A) followed by the same single dose under fed conditions (treatment B).
  Interventions: Drug: CANA/MET XR FDC
- Sequence BA (Experimental): A single dose of CANA/MET XR FDC tablet of 150 mg/1,000 mg under fed conditions (treatment B) followed by the same single dose under fasted conditions (treatment A).
  Interventions: Drug: CANA/MET XR FDC

INTERVENTIONS:
Drug: CANA/MET XR FDC — Canagliflozin/extended release Metformin (CANA/MET XR) fixed dose combination (FDC) tablet of 150 mg/1,000 mg

SUMMARY:
The purpose of this study is to assess the effect of coadministration of a high-fat meal on the oral bioavailability of a fixed dose combination of Canagliflozin/extended release Metformin (CANA/MET XR) tablet, containing 150 mg CANA and 1,000 mg extended release MET in healthy participants.

DETAILED DESCRIPTION:
This is a randomized (a sequence of fasted and fed periods accompanying study drug intake will be assigned by chance), open-label (physicians and participants know the identity of the assigned treatment), single-center, single-dose, 2-period, 2-sequence, crossover study of Canagliflozin/extended release Metformin (CANA/MET XR) fixed dose combination (FDC) tablet of 150 mg/1,000 mg. Approximately 24 healthy adult participants will be enrolled to ensure that at least 20 complete the study.

After a screening period, participants will be randomly assigned to 1 of the 2 treatment sequences (AB or BA) on Day 1 of Period 1. Treatment A means a participant will receive a single 150/1,000 mg CANA/MET XR FDC tablet under fasted conditions, and Treatment B means that a participant will receive the same drug under fed conditions. Participants will need to remain at the study center for 4 days (72 hours postdose) after the drug administration for collection of blood samples in each treatment period. There will be a 10- to 14-day washout period between Period 1 and Period 2. On Day 4 (72 hours postdose) of Period 2, when participants are discharged from the study center, they will be given instructions to return for a follow-up visit 7 to 10 days later. For Treatment B (in fed state), participants will be provided with a standardized high-fat breakfast. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent document indicating they understand the purpose of the study and procedures
* Must have a body mass index (BMI) of between 18 and 30 kg/m², inclusive
* Must have a body weight of not less than 50 kg
* Must have a blood pressure between 90 and 140 mmHg inclusive, systolic, and no higher than 90 mmHg diastolic at screening
* Must have normal renal function and no evidence of kidney damage (including abnormalities in blood or urine tests)

Exclusion Criteria:

* History of or current clinically significant medical illness
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements)
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose- Known allergy to heparin or history of heparin induced thrombocytopenia
* History of smoking or use of nicotine-containing substances within the previous 2 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of canagliflozin following the single dose of CANA/MET XR FDC after fed and fasted conditions | Predose, (before tablet intake) up to 72 hours afterdose
  Plasma concentrations of canagliflozin are used to evaluate how long canagliflozin stays in the body.
Plasma concentration of metformin following the single dose of CANA/MET XR FDC after fed and fasted conditions | Predose, up to 72 hours afterdose
  Plasma concentrations of metformin are used to evaluate how long metformin stays in the body.

SECONDARY OUTCOMES:
Percentage of participants with adverse events as a measure of safety and tolerability | Screening, up to Day 10 of the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Lincoln, Nebraska, United States